CLINICAL TRIAL: NCT02420132
Title: Decentralized Pilot Study to Evaluate MyVisionTrack^TM Home Vision Testing in Patients With Diabetic Macular Edema or Neovascular Age-Related Macular Degeneration Currently Receiving Intravitreal Lucentis® Therapy.
Brief Title: Study to Evaluate Home Vision Testing in Participants Who Receive Ranibizumab (Lucentis®)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: GE29720
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Macular Edema; Macular Degeneration
MeSH Terms: conditions — Macular Edema; Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Main Study: Decentralized participant recruitment, participant and local ophthalmologist compliance, and use of the mVT mobile medical application in a more geographically diverse, decentralized cohort of participants with DME or nAMD receiving intravitreal ranibizumab therapy as part of standard-of-care treatment.
  Interventions: Other: Ranibizumab
- Traditional Substudy: Subset of participants enrolled through a single investigator who will determine visual acuity and anatomical markers of disease status using clinical "gold standard" assessments (certified ETDRS protocol visual acuity and macula OCT).
  Interventions: Other: Ranibizumab

INTERVENTIONS:
Other: Ranibizumab — Ranibizumab administered as part of standard-of-care

SUMMARY:
This pilot study will evaluate home vision testing using a mobile medical application in participants with diabetic macular edema (DME) or neovascular age-related macula degeneration (nAMD) who receive intravitreal ranibizumab therapy. In the main, decentralized study, participants will be recruited via digital media, advocacy groups, or through their own ophthalmologist. The traditional substudy will evaluate the association between visual acuity and anatomical markers of disease status determined using clinical "gold standard" assessments (certified Early Treatment Diabetic Retinopathy Study [ETDRS] protocol visual acuity and macula optical coherence tomography [OCT]) and the results of home vision testing using the myVisionTrack^TM (mVT) application.

ELIGIBILITY:
Inclusion Criteria:

* DME or active nAMD in at least one eye
* Current treatment with intravitreal ranibizumab therapy, with evaluations planned every 4 to 8 weeks
* Access to an approved mobile device with a data plan or WiFi internet access

Exclusion Criteria:

* Any other eye condition causing eye disease that limits vision and cannot be corrected, other than DME or nAMD
* Dementia or other neurologic or psychological limitation that would prevent the participant from performing regular self-testing of visual function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who are receiving treatment for DME or nAMD with intravitreal ranibizumab and are being evaluated at intervals of 4-8 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2016-08-25 (Actual)

PRIMARY OUTCOMES:
Number of "Clicks" on Study Information Advertisements on Participant Advocacy, Digital Media, and Professional Society Websites (Main Study Only) | Baseline up to 6 months
Percentage of Participants Participating at Specified Milestones in the Recruitment/Enrollment Process (Main Study Only) | Baseline up to 6 months
Percentage of Participants Performing Self-Testing Two Times per Week Using the Mobile Medical Application | Baseline up to 6 months
Percentage of Participants Visiting their Ophthalmologist at Least Every 8 Weeks (Main Study Only) | Baseline up to 6 months
Percentage of Office Visits for which Visual Acuity Data Were Provided to Scripps Translational Science Institute (STSI) (Main Study Only) | Baseline up to 6 months
Percentage of Office Visits for which OCT Data Were Provided to STSI (Main Study Only) | Baseline up to 6 months
Degree of Correlation Between mVT Test Results and Certified ETDRS Protocol Visual Acuity (Traditional Substudy Only) | Baseline up to 6 months
Degree of Correlation between mVT Test Results and OCT Characteristics (Traditional Substudy Only) | Baseline up to 6 months

SECONDARY OUTCOMES:
Association Between mVT Test Results and Routine Visual Acuity Measurements, Measured by Snellen or Other Standard-of-Care Visual Acuity Scores (Main Study Only) | Baseline up to 6 months
Total Number of Participants in the Enrolled Population (Main Study Only) | Baseline up to 6 months
Total Number of Participants in the Confirmed Population (Main Study Only) | Baseline up to 6 months
Differences Between the Participant's and their Ophthalmologist's Assessments of Eligibility (Main Study Only) | Baseline up to 6 months
Percentage of Photographed and Transmitted OCT Images that Are Gradable for Central Subfield Thickness | Baseline up to 6 months
Percentage of Participants Downloading the mVT Application who Require Assistance via Human Interaction from the Help Lines | Baseline
Number of Support Tickets Needed for Technician/Coordinator Interactions with the Participant to Download the mVT Application | Baseline
Total Support Time as an Average per Participant Needed for Technician/Coordinator Interactions with the Participant to Download the mVT Application | Baseline
Number of Additional Support (Calls/Interactions) Required by Participants | Baseline up to 6 months
Number of Critical Security Issues which May Require Reporting | Baseline up to 6 months
Number of Losses of Participant Data Due to Technical Issues | Baseline up to 6 months
Number of Data Processing Issues Occurring During the Study that Are Recoverable but Require Specific Effort, Indicating a Technical Problem | Baseline up to 6 months
Score of Participants Survey on Opinions Regarding Self-Monitoring | At 1 week and 3 months after enrollment, at study completion/participant withdrawal (up to 6 months)
Percentages of Substudy OCT Images (Photographs of the OCT Taken Using a Mobile Device), that Are Readable for Qualitative Assessment, Readable for Quantitative Assessment, or Indeterminate (Traditional Substudy Only) | Baseline up to 6 months
Percentage of Actual Substudy Downloaded OCT Images that Are Readable for the Presence of Cysts, Sub Retinal Fluid, and Pigment Epithelial Detachment, or Indeterminate (Traditional Substudy Only) | Baseline up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Rocky Mountain Retina, Salt Lake City, Utah, United States